CLINICAL TRIAL: NCT06503029
Title: Cytotoxicity, Leaching, and Structural Conformation of Invisalign Clear Aligners Subjected to Different Cleaning Methods: A Randomized Controlled Trial
Brief Title: Evaluate Cytotoxicity, Leaching, and Structural Conformation of Clear Aligners
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Yara AlSenani, Resident, Riyadh Elm University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FPGRP/2024/823/1114
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Malocclusion; Cytotoxicity
Keywords: Cytotoxicity; Leaching; Clear aligner; Orthodontics
MeSH Terms: conditions — Malocclusion | interventions — Hydrotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: To maintain anonymity, unique identification numbers will be generated for each patient, and the data obtained will be carefully coded. This will ensure that patient data is kept separate from other collected data and stored in a secure and protected location.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Invisalign Cleaning Crystals (Experimental): Invisalign Cleaning Crystals are used as a cleaning method for orthodontic clear aligners. It includes Sodium Sulfate as an active ingredient.
  Interventions: Device: Invisalign Cleaning Crystals
- Fittey Dent Cleaning Tablet (Experimental): Fittey Dent Cleaning Tablet is used as a cleaning method for orthodontic clear aligners. It includes Sodium Perborate as an active ingredient.
  Interventions: Device: Fittey Dent Cleaning Tablet
- Listeren Mouthwash used as cleaning method (Experimental): Listeren Mouthwash is used as a cleaning method for orthodontic clear aligners. It includes Eucalyptol and Menthol as active ingredients.
  Interventions: Drug: Listeren Mouthwash
- Toothbrush and water (Active Comparator): Toothbrush and water is used as a cleaning method for orthodontic clear aligners that as recommended by the aligner manufacturer.
  Interventions: Device: Toothbrush and Water

INTERVENTIONS:
Device: Invisalign Cleaning Crystals — Invisalign Cleaning Crystals are used as a cleaning method for orthodontic clear aligners. It includes Sodium Sulfate as an active ingredient.
  Arms: Invisalign Cleaning Crystals
Device: Fittey Dent Cleaning Tablet — Fittey Dent Cleaning Tablet is used as a cleaning method for orthodontic clear aligners. It includes Sodium Perborate as an active ingredient.
  Arms: Fittey Dent Cleaning Tablet
Drug: Listeren Mouthwash — Listeren Mouthwash is used as a cleaning method for orthodontic clear aligners. It includes Eucalyptol and Menthol as active ingredients.
  Arms: Listeren Mouthwash used as cleaning method
Device: Toothbrush and Water — Toothbrush and water is used as a cleaning method for orthodontic clear aligners that as recommended by the aligner manufacturer.
  Arms: Toothbrush and water

SUMMARY:
The aim is to evaluate clear aligners' cytotoxicity, leaching, and structural properties and compare them with four cleaning tools. The null hypothesis is the cleansers have no impact on the properties tested.

DETAILED DESCRIPTION:
Orthodontic Invisalign clear aligners patients will be randomly distributed into four groups using four cleaning methods. Participants will be instructed to clean their trays as instructed by the production company.

Leaching, Cytotoxicity, and Structural Confirmation will be evaluated of the Invisalign clear aligners after being used.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are on Invisalign Clear aligner treatment.
* Participants who are 21 years and older and committed to their treatment.
* Participants with caries-free dentition
* Participants with no smoking habits
* Participants are not pregnant females

Exclusion Criteria:

* Participants who are on Orthognathic treatment.
* Participants with Hypodontia.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-01-25 (Estimated); Study Completion 2025-03-05 (Estimated)

PRIMARY OUTCOMES:
Cytotoxicity | 1-2month
  Aligners from each of the four groups will be submerged in normal saline for a month at 37°C to conduct a cytotoxicity assessment. Following that, the solutions were diluted to three distinct concentrations (5%, 10%, and 20% volume/volume). After 48 hours of seeding in 96-well microplates, gingival fibroblasts were exposed to the solution, and the medium will be changed to an MTT solution (MTT: 3-[4,5-dime-thylthiazol-2-yl]-2,5-diphenyltetrazolium bromide). Then optical density will be measured to ascertain cell viability and subsequently assess cytotoxicity.
Leaching | 1-2months
  Each set of aligners from each of the four groups will be cut into 5x5 mm squares. To accelerate the degradation of the sample, each specimen will be submerged in a single glass vial with an alcoholic media. Each material will be soaked in five different solutions as follows: the first is absolute ethanol (100%), the second is 75% ethanol to 25% water, the third is 50% ethanol to water, the fourth is 25% ethanol to 75% water, and finally, 100% water solution served as the control.
  A gas chromatography-mass spectrometry unit shall be used to analyze the leached substances in the immersion medium. An Agilent GC 7890A combined with a triple-axis detector 5975 C single quadrupole mass spectrometer will be used for GC-MS analysis
Structural Conformation | 1-2months
  Maxillary and mandibular clear aligners from all four included groups will be cut into 5 × 5 mm squares. Each specimen will be mounted in a plastic mold using an orthodontic plaster to facilitate the indentation process. The microhardness will be tested using a Vickers indenter (INNOVATEST, FALCON 450, Deutschland GmbH) by applying a 25 gf load for 15 s.

CONTACTS AND LOCATIONS:
Overall Officials: Omar AlKadhi, BDS,MSc, Principal Investigator — Associated Professor, Riyadh Elm University.
Locations (1):
- Riyadh Elm University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahrari F, Tavakkol Afshari J, Poosti M, Brook A. Cytotoxicity of orthodontic bonding adhesive resins on human oral fibroblasts. Eur J Orthod. 2010 Dec;32(6):688-92. doi: 10.1093/ejo/cjq019. Epub 2010 Jun 21. PMID 20570954
- [Background] Alhendi A, Khounganian R, Almudhi A. Cytotoxicity assessment of different clear aligner systems: An in vitro study. Angle Orthod. 2022 Sep 1;92(5):655-660. doi: 10.2319/121621-919.1. Epub 2022 Jun 7. PMID 35666210
- [Background] Alhendi A, Khounganian R, Almudhi A, Ahamad SR. Leaching of Different Clear Aligner Systems: An In Vitro Study. Dent J (Basel). 2022 Feb 14;10(2):27. doi: 10.3390/dj10020027. PMID 35200252
- [Background] Eliades T, Pratsinis H, Athanasiou AE, Eliades G, Kletsas D. Cytotoxicity and estrogenicity of Invisalign appliances. Am J Orthod Dentofacial Orthop. 2009 Jul;136(1):100-3. doi: 10.1016/j.ajodo.2009.03.006. PMID 19577155